CLINICAL TRIAL: NCT00005922
Title: Role of Conditioning in the Pharmacotherapy of Psoriasis
Brief Title: Conditioning, the Placebo Effect, and Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Robert Ader, Ph.D., University of Rochester School of Medicine and Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AR046825 (NIH); R01AR046825 (NIH); NIAMS-051
Record Dates: First submitted 2000-06-22; First posted 2000-06-23 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Psoriasis
Keywords: Conditioning; Corticosteroid; Lesions; Pharmacotherapy; Placebo effect; Psoriasis; Psychoneuroimmunology
MeSH Terms: conditions — Psoriasis | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Participants will receive 100% of the dose of the medication on the same reinforcement schedule (100%) as received during the baseline (maintenance) period.
  Interventions: Other: Standard pharmacotherapeutic protocol
- B (Experimental): Participants will receive 100% of the dose of the medication on a partial reinforcement schedule (25% or 50%) as received during the baseline (maintenance) period
  Interventions: Behavioral: Partial schedule of pharmacotherapeutic reinforcement
- C (Experimental): Participants will receive 25% or 50% of the dose of the medication on the same reinforcement schedule (100%) as received during the baseline (maintenance) period.
  Interventions: Drug: Dose control for Arm B

INTERVENTIONS:
Behavioral: Partial schedule of pharmacotherapeutic reinforcement — Dose of 0.1% of Aristocort A on 1-2 of every 4 days for a period of up to 14 weeks.
  Other Names: Aristocort A
  Arms: B
Drug: Dose control for Arm B — Dose of 0.025-0.05% of Aristocort A 2 times per day for a period of up to 14 weeks.
  Other Names: Aristocort A
  Arms: C
Other: Standard pharmacotherapeutic protocol — Full dose of Aristicort A (0.1%) 2 times per day for a period of up to 14 weeks.
  Other Names: Aristicort A
  Arms: A

SUMMARY:
This study uses the psychological principle known as classical conditioning to try to improve the standard treatment of psoriasis. Classical conditioning is a process of behavioral modification in which a person learns to connect a certain response-in this case, improvement of psoriasis-with a new action, or stimulus-in this case, application of an inactive cream. The goal of this study is to show that people with psoriasis who are maintained on corticosteroid cream part of the time and an inactive (placebo) cream at other times show a lower incidence of relapse and a reduced severity of psoriasis that patients treated with that same (reduced) amount of medication administered all the time.

DETAILED DESCRIPTION:
The lack of scientific attention devoted to the placebo effect as a phenomenon in its own right probably reflects the paucity of theoretical positions within which to organize the existing data and design new research. This research addresses the clinical significance of behavior-immune system interactions.

This study will capitalize on conditioned immunosuppressive responses to reduce the cumulative amount of corticosteroid medication used in the treatment of psoriasis. We will continue to treat patients with steroid, but will shift experimental patients from their current schedule of continuous reinforcement (active drug whenever medication is applied) to a partial schedule of reinforcement (active drug a percentage of the time and placebo alone at other times). To equate amount of medication, we will treat another group of patients with a reduced dose of steroid in a standard treatment regimen (continuous schedule of reinforcement).

We hypothesize that, holding cumulative dose constant, a partial schedule of reinforcement will enable patients to be maintained on lower cumulative amounts of corticosteroid than patients treated under a continuous schedule of active drug. This is the first attempt to adopt conditioning principles and use schedules of reinforcement to design regimens of drug therapy. If proven effective, this new approach to pharmacotherapy and placebo effects is likely to stimulate new interdisciplinary research in neuropharmacology and behavioral pharmacology for the treatment of autoimmune disorders and a variety of other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis patients with mild to moderate lesions who are able to attend weekly clinic visits at either the University of Rochester School of Medicine and Dentistry in Rochester, NY, or Stanford University in Palo Alto, CA.
* Patients must be in good health (as determined by prescreening examination).
* Patients must not be using systemic treatment (for example, oral medications) or intralesional, UV, or topical therapies except bland emollients for at least 2 weeks before the start date of the study.
* Patients must have chronic, stable plaque psoriasis with a score of greater than or equal to 7 on a routine 9-point Severity Index.

Exclusion Criteria:

* Use of immunosuppressive medication within the past 2 months.
* Pregnant or sexually active women who do not use contraceptives.
* Patients who cannot be monitored regularly.
* History of allergy to corticosteroid or other study ointment components.
* Patients who have more than 10 percent of body surface area covered by psoriatic lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2000-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Routine and standard quantitative and qualitative assessment of plaque changes and growth | Weekly
Severity Index, clinically described as to redness, flaking and thickness on a total scale of 9 | Weekly

SECONDARY OUTCOMES:
Impacts of Events Scale (IES) | Once - at the initial start of the study
Psoriasis Life Stress Inventory) (PLSI) | Weekly
Hassles Scale | Weekly
Interpersonal Support Evaluation List (ISEL) | Once - at the intial start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ader, PhD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Adult Dermatology Clinic, Strong Memorial Hospital, Rochester, New York

REFERENCES:
- [Background] Ader R, Cohen N. Behaviorally conditioned immunosuppression. Psychosom Med. 1975 Jul-Aug;37(4):333-40. doi: 10.1097/00006842-197507000-00007. PMID 1162023
- [Background] Ader R, Cohen N, Felten D. Psychoneuroimmunology: interactions between the nervous system and the immune system. Lancet. 1995 Jan 14;345(8942):99-103. doi: 10.1016/s0140-6736(95)90066-7. No abstract available. PMID 7815892
- [Background] Giang DW, Goodman AD, Schiffer RB, Mattson DH, Petrie M, Cohen N, Ader R. Conditioning of cyclophosphamide-induced leukopenia in humans. J Neuropsychiatry Clin Neurosci. 1996 Spring;8(2):194-201. doi: 10.1176/jnp.8.2.194. PMID 9081556
- [Background] Ader R. "The role of conditioning in pharmacotherapy." In The placebo effect: An interdisciplinary exploration, edited by A. Harrington, 138-165. Cambridge: Harvard University Press, 1997.